CLINICAL TRIAL: NCT02905552
Title: Myelodysplasic Syndromes and Risk Factors for Infection : A Case / Control Study
Brief Title: Myelodysplasic Syndromes and Risk Factors for Infection
Acronym: MYRIFIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI13004
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Myelodysplastic Syndrome (MDS); Infection; Risk Factors; IPSS High Risk
Keywords: Myelodysplastic syndrome (myelodysplasia); Infection; Risk Factors
MeSH Terms: conditions — Myelodysplastic Syndromes; Infections; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case group: Patient developing a first episode of infection since diagnosis of high-risk MDS (index case)
  Interventions: Other: No intervention
- Control group: Patient with no infection since diagnosis of MDS
  Patient will be paired to index case by:
  * Hospital site
  * Age
  * Sexe Control patient is eligible if he has been seen in consultation within 15days before or after date of first infection of index case If matching fails, control patient can be found in another site and/or within 30days before or after date of first infection of index case
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Myelodysplastic Syndromes (MDS) are characterized by quantitative and qualitative bone marrow failure and by a disorder of the medullary production which is a pre-leukemic state which can evolve into acute myeloid leukemia.

The risk of leukemic transformation is estimated by the score IPSS (International Prognostic Score System). We distinguish the MDS of low risk (IPSS<1) and those of high risk of leukemic transformation (IPSS=1,5).

Besides the risk of leukemic transformation, MDS much be complicated of infections which could be life-threatening.

The risk of developing first infection after the diagnosis of MDS of high risk is probably influenced by anamnestic (disease duration, comorbidities), clinical (veinous central catheter, previous hospitalization), biological (neutropenia, lymphopenia, serum ferritin) and therapeutics (demethylating agent, lenalidomide, erythropoietin, G-CSF, transfusions, anti-infectious preventive treatment) factors. Their identification will allow for improved targeting of the population which is is likely to benefit from anti-infective prophylaxis Primary objective is to identify risk factors associated with first acute episode of infection in patients with MDS, by comparing index cases and matched control cases who did not develop infection episode since diagnosis.

Secondary objectives are to explore nature and severity of infectious episodes, number of recurrences during 1 year of follow up and survival at 6 and 12 months

DETAILED DESCRIPTION:
* 160 couples (Case / Control)
* Pairing according to age (+/- 5 years), sex and medical consultation date (+/-15 days)
* Follow up at M3, M6, M9 and M12
* Study duration : 24 months
* Inclusion duration : 12 months

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* MDS with IPSS >1.5
* With a first infectious episode since the diagnosis of SMD of high risk (Case)
* Unhurt of any infection and being able to be mated in the case index (Control)
* Consulting or hospitalized in one of the services involved in the study during the period of inclusion

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-risk MDS (IPSS > 1,5)
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of infectious episode | 12 months follow-up

SECONDARY OUTCOMES:
severity of infectious episode | 12 months follow-up
Overall Survival (all-cause mortality) | 12months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Toma, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France